CLINICAL TRIAL: NCT02711228
Title: Study of Immune Deficiency Patients Treated With Subcutaneous Immunoglobulin (IgPro20, Hizentra®) on Weekly and Biweekly Schedules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IgPro20_4005; 2015-004977-34 (EudraCT Number)
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Primary Immune Deficiency; Secondary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subcutaneous Immune Globulin (Human) (Hizentra) (Experimental): Hizentra, Subcutaneous Immune Globulin (Human) (SCIg), is a ready to use, polyvalent human normal Immunoglobulin G (IgG) for subcutaneous administration. Hizentra is a 20% IgG protein solution, is prepared from large pools of human plasma, and is stabilized by L-Proline.
  Interventions: Biological: Subcutaneous Immune Globulin (Human) (Hizentra)

INTERVENTIONS:
Biological: Subcutaneous Immune Globulin (Human) (Hizentra) — Hizentra, Subcutaneous Immune Globulin (Human) (SCIg), is a ready to use, polyvalent human normal Immunoglobulin G (IgG) for subcutaneous administration. Hizentra is a 20% IgG protein solution, is prepared from large pools of human plasma, and is stabilized by L-Proline.
  Other Names: IgPro20; Hizentra

SUMMARY:
The purpose of the study is to assess the impact of immunoglobulin treatment by subcutaneous injections every 2 weeks (biweekly) on a cohort of patients with primary and secondary immune deficiencies. The full study will consist of safety, efficacy and Quality of Life (QoL) evaluations and a pharmacokinetic (PK) sub-study. The primary objectives of the study are to determine tolerability and safety of biweekly IgPro20 injection regimen and to compare PK outcomes on weekly and biweekly IgPro20 therapy.

Patients who have received and/or are currently receiving immunoglobulin G (IgG) in intravenous (IVIg), or subcutaneous (SCIg) infusions are eligible for inclusion if they meet inclusion/exclusion criteria.

The study consists of two parts. In Part 1 of the study enrolled subjects will receive IgPro20 weekly for either 12 weeks (for patients on SCIg infusion prior to the study) or 24 weeks (for patients on IVIg infusion prior to the study). Part 2 will consist of a biweekly treatment with IgPro20 for 52 weeks, for both groups.

Additionally, study subjects meeting inclusion criteria for the PK sub-study will undergo a PK sample collection for 1 week and 2 weeks in study Parts 1 and 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

Full study:

* Female or male patients with primary or secondary immunodeficiency, aged from 5 to 64 years, receiving steady state immunoglobulin G replacement therapy.

Pharmacokinetic sub-study:

* Female or male patients with primary immunodeficiency, aged between 12 and 64 years of age, on steady-state IgPro20 replacement therapy and willing to undergo pharmacokinetic sample collection on weekly and biweekly IgPro20 dosing regimens.

Exclusion Criteria:

* Patients with protein losing conditions such as: lymphangiectasis, nephrosis, status post cardio-thoracic surgery requiring drainage tubes for more than 48 hours, protein-losing enteropathy.
* Concomitant treatment with plasma or other blood products (including any IgGs other than IgPro20 [Hizentra]) within 21 days before study entry and/or during the study.
* Any other condition or treatment that, in the opinion of the investigator, would interfere with obtaining valid results for that subject.
* Women of childbearing potential with a positive pregnancy test.
* Active infection at the time of screening.

Ages: 5 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Annualized rate of adverse events (local and systemic) | During biweekly treatment period, up to approximately 52 weeks
Area under the concentration-time curve, AUC(0-t ) | Immediately before, and up to 7 days after infusion during the weekly treatment period and up to 14 days after infusion during the biweekly treatment periods.
Maximal serum IgG concentration (Cmax) | Up to 7 days after infusion during the weekly treatment period and up to 14 days after infusion during the biweekly treatment periods.
Time to maximal serum IgG concentration (Tmax) | Up to 7 days after infusion during the weekly treatment period and up to 14 days after infusion during the biweekly treatment periods.
Trough serum IgG concentration (Ctrough) | Immediately before, and up to 7 days after infusion during the weekly treatment period and up to 14 days after infusion during the biweekly treatment periods.

SECONDARY OUTCOMES:
Annualized rate of infections per patient | During weekly and biweekly treatment periods, up to approximately 64 - 76 weeks
Serum IgG trough levels (Ctrough) | On day 7 (immediately before each next infusion) during the weekly treatment period, and on week 24 and 48 of biweekly treatment.
Health-related Quality of Life | During weekly and biweekly treatment periods, up to approximately 64 - 76 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elie Haddad, MD, Principal Investigator — St. Justine's Hospital
Locations (2):
- Canada (2):
  - Centre Hospitalier de l'université de Montréal, Montreal
  - CHU Sainte-Justine, Montreal

IPD SHARING:
Plan to Share IPD: Undecided